CLINICAL TRIAL: NCT04752150
Title: Comparison of Ultrasound-Guided Erector Spinae Plane Block and Rhomboid Intercostal Block for Pain Management Following Mastectomy Surgery
Brief Title: ESPB and RIB for Pain Management Following Mastectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 18
Record Dates: First submitted 2021-02-01; First posted 2021-02-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female
Keywords: Mastectomy and axillary dissection surgery; Postoperative pain management; Rhomboid intercostal block; Erector spina plane block
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is ESPB group. The second one is RIB group
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation and the patient will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB = Erector spinae plane block group (Active Comparator): In group ESPB, ESPB will be performed with patients in the lateral decubitus position while the surgical site up. US probe will be placed 2-3 cm lateral to the T4 transvers process. The block needle will be inserted cranio-caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 30 ml %0.25 bupivacaine will be administered for block.
  Interventions: Other: Analgesia management; group ESPB and RIB
- Group RIB = RIB group (Active Comparator): In group RIB, RIB block will be performed with patients in the lateral decubitus position while the surgical site up. The linear high frequency probe will be placed in sagittal plane medially on the medial border of the scapula at T5-6 level. The trapezius muscle, rhomboid major muscle, intercostal muscle, ribs and the pleura will be visualized. The needle will be inserted into the fascial plane between the rhomboid major and intercostal muscles in a cranio-caudal direction. A dose of 30 ml 0,25% bupivacaine will be injectted into the fascial plane.
  Interventions: Other: Analgesia management; group ESPB and RIB

INTERVENTIONS:
Other: Analgesia management; group ESPB and RIB — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Postoperative pain is an important issue in patients underwent mastectomy and axillary dissection surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay. The US-guided erector spina plane block (ESPB) may be used for postoperative pain treatment following breast surgery. It is a novel interfascial block that was defined by Forero. Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. Local anesthetic solution is administrated between the rhomboid muscle and intercostal muscles over the T5-6 ribs. It has been reported that RIB may provide effective analgesia management for several breast surgeries.

The primary aim of the study is to compare postoperative pain scores (VAS), and the secondary aim is to evaluate postoperative opioid consumption, adverse effects related with opioids (allergic reaction, nausea, vomiting).

DETAILED DESCRIPTION:
Postoperative pain is an important issue in patients underwent mastectomy and axillary dissection surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following mastectomy and axillary dissection surgery. Ultrasound (US)-guided interfascial plane blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice. Rhomboid intercostal block (RIB) is a novel block and was first described by Elsharkawy et al. Local anesthetic solution is administrated between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2-3 cm medially of the medial border of the scapula. RIB targets both the posterior rami and lateral cutaneous branches of the thoracic nerves and provides analgesia for the hemithorax from T2 to T9. It has been reported that RIB may provide effective analgesia management for several breast surgeries.

The US-guided erector spina plane block (ESPB) is defined by Forero et al. ESPB provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. ESPB contains a local anesthetic injection into the deep fascia of erector spinae. Visualization of sonoanatomy is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. In the literature, it has been reported that ESP block provides effective analgesia after several surgeries such as open heart surgery, breast surgery, thoracoscopic and abdominal operations.

The aim of this study is to evaluate the efficacy of the US-guided ESPB and RIB for postoperative analgesia after mastectomy and axillary dissection surgery. The primary aim is to compare postoperative pain scores (VAS), and the secondary aim is to evaluate opioid consumption, adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for mastectomy and axillary dissection surgery under general anesthesia

Exclusion Criteria:

* receiving anticoagulant treatment,
* known study drugs allergy,
* opioid addiction
* infection of the skin at the site of the block,
* pregnancy or lactation,

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who will undergo breast surgery will be included
Enrollment: 60 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16, and 24 hours.
  The primary aim is to compare VAS. Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded

SECONDARY OUTCOMES:
Opioid consumption | Change from baseline opioid consumption at postoperative 1, 2, 4, 8, 16, and 24 hours
  The secondary aim is to compare postoperative opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Ciftci B, Ekinci M, Celik EC, Tukac IC, Bayrak Y, Atalay YO. Efficacy of an Ultrasound-Guided Erector Spinae Plane Block for Postoperative Analgesia Management After Video-Assisted Thoracic Surgery: A Prospective Randomized Study. J Cardiothorac Vasc Anesth. 2020 Feb;34(2):444-449. doi: 10.1053/j.jvca.2019.04.026. Epub 2019 Apr 30. PMID 31122843
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Dere O, Ugur B. Evaluation of ultrasound-guided rhomboid intercostal nerve block for postoperative analgesia in breast cancer surgery: a prospective, randomized controlled trial. Reg Anesth Pain Med. 2020 Apr;45(4):277-282. doi: 10.1136/rapm-2019-101114. Epub 2020 Feb 19. PMID 32079739